CLINICAL TRIAL: NCT02604277
Title: Suicidal Behavior in Patients Diagnosed With Bipolar Disorder: The Roles of Biological and Childhood and Adult Environmental Risk Factors
Brief Title: Suicidal Behavior in Patients Diagnosed With Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Dorian Lamis, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00084800; 2025P010887 (Other: Emory IRB)
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Depression; Alcoholism; Drug Abuse
Keywords: Psychology
MeSH Terms: conditions — Depression; Alcoholism; Substance-Related Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Intervention Program (Experimental): Patients diagnosed with Bipolar Disorder will receive therapy in a group setting of 4 to 12 male and female participants.
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy (ISRT); Behavioral: Bipolar-Specific Cognitive Behavioral Therapy (CBT); Behavioral: Mindfulness-Based Stress Reduction (MBSR); Behavioral: Psycho-education & Understanding Bipolar Medications Therapy

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy (ISRT) — Interpersonal and Social Rhythm Therapy (ISRT) will be given once a week over a six week period for 55-60 minutes. ISRT emphasizes identifying and maintaining a regular routine in daily life. It includes addressing sleep and solving interpersonal concerns and conflicts by focusing on daily routine.
Behavioral: Bipolar-Specific Cognitive Behavioral Therapy (CBT) — Bipolar-Specific Cognitive Behavioral Therapy (CBT) will be given once a week over a six week period for 55-60 minutes.The therapy is directly focused on eliminating or managing specific problems experienced by people with Bipolar Disorder. As part of this intervention, participant's maladaptive thoughts, behaviors and emotions are identified followed by learning how to challenge negative thoughts and reframing into positive, more adaptive thoughts. Additionally, the intervention involves enhancing the participant's coping skills and the ability to view a situation more objectively.
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Mindfulness-Based Stress Reduction (MBSR) will be given once a week over a six week period for 55-60 minutes. MBSR is a structured intervention that utilizes mindfulness meditation to reduce suffering associated with physical and psychiatric illnesses. MBSR is nonreligious in nature and aims to encourage an enhanced awareness of moment-to-moment experience of noticeable mental processes.
Behavioral: Psycho-education & Understanding Bipolar Medications Therapy — Psycho-education & Understanding Bipolar Medications Therapy will be given once a week over a six week period for 55-60 minutes. Psycho-education & Understanding Bipolar Medications Therapy aims to provide psycho-education about Bipolar Depression as well as provide a platform for participants to address concerns about managing their illness. Issues such as managing symptoms, reducing relapses and hospitalizations as well as maintaining gains will be discussed

SUMMARY:
The purpose of this study is to learn the environmental and psychological factors that impact suicidality in patients diagnosed with Bipolar Disorder. Additionally, the study aims to identify treatments to reduce the suicidal behavior and improve quality of life through a 6-week group-based intervention program.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a severe, chronic, and relatively common psychiatric illness associated with significant premature mortality, including death by suicide. Given that suicidal behavior is a major public health problem and BD confers the highest risk of suicide among major mental disorders, it is important for clinical researchers to investigate why individuals with BD are at an increased risk for suicidal thoughts and behaviors. Among those diagnosed with BD, approximately 75% of patients experience suicidal ideation in their lifetime, 30% attempt suicide, and about 20% eventually die by suicide. Research has also demonstrated that suicidal acts in BD patients tend to be more lethal as indicated by a lower ratio of attempted suicide to death than in the general population. Given that BD patients use more dangerous suicide methods and die by suicide at an alarmingly high rate, early identification and appropriate treatment are critical. Thus, the proposed study should provide critical information and inform treatment efforts regarding suicide risk in low income BD patients.

Research has consistently demonstrated that childhood maltreatment, including abuse and neglect, are independently associated with increased risk for suicidal ideation/behavior in a variety of populations, including patients diagnosed with BD. Consequently, inquiring about past childhood abuse and neglect when assessing suicide risk in this vulnerable population is important. Moreover, childhood maltreatment has been shown to contribute to impulsive aggression and adult drug use, both of which have been shown to predict suicidal behavior in BD patients. Castroman and colleagues (2014) demonstrated that impulsive aggression was an intermediate factor linking childhood abuse with the severity of suicidal behavior in a large sample of suicide attempters. Similarly, Roy (2011) found that impulsive aggression was a significant mediator in the association between childhood abuse and suicidal behavior in substance-dependent patients. With regards to substance use, current evidence suggests that among individuals abused in childhood, the risk for drug use and subsequent suicidal behavior is increased. Further, among BD patients in particular, there appears to be significant additive effects of childhood maltreatment and drug abuse on suicide attempts.

The associations among these variables may be best explained by the interpersonal-psychological theory of suicide (IPTS), which provides a conceptual framework for understanding why individuals consider and engage in suicidal behavior. The theory differentiates between the desire for suicide and the capability of engaging in suicide behaviors among suicide attempters. Desire is characterized by two constructs, perceived burdensomeness (i.e., one's death is worth more than one's life to others) and thwarted belongingness (i.e., sense of alienation and disconnection). Suicide attempts and deaths are arguably related to the ability to use lethal means on one's self, and require pain tolerance and a developed sense of fearlessness in the face of death. Specifically, Joiner (2005) posits that the capability to initiate suicidal behavior is acquired via exposure to painful and fear-provoking events (e. g., childhood maltreatment) that habituate individuals to the pain and fear associated with death. Consequently, understanding pathways by which distal factors, such as childhood maltreatment, may influence suicidal capability is crucial. The proposed investigation of potential developmental pathways from childhood maltreatment to suicidal behaviors through the risk factors of impulsive aggression and drug use may elucidate the associations among these variables, and subsequently improve the assessment and treatment of suicidal BD patients. Thus, the proposed investigation will focus on the capability to engage in suicidal behaviors as examining all ITPS constructs is beyond the scope of this study. More specifically, the researchers propose to examine the relationships between these environmental and psychological factors in BP patients.

The purpose of this study is to learn the environmental and psychological factors that impact suicidality in patients with Bipolar Disorder. Additionally, the study aims to identify treatments to reduce the suicidal behavior and improve quality of life through a 6-week group-based intervention program. Groups will include topics such as interpersonal/social rhythm and mindfulness interventions, as well as interventions focused on understanding and changing thoughts to better cope with Bipolar Depression.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of Bipolar Disorder (BD)
* Able to provide written informed consent

Exclusion Criteria:

* Cognitive impairments
* Acutely psychotic
* Medically unstable
* History of schizophrenia spectrum disorder
* History of mood incongruent psychotic symptoms
* History of primary substance disorder
* History of primary organic disease and/or dementia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Pre-intervention, Post-intervention (Up to six weeks)
  Columbia-Suicide Severity Rating Scale (C-SSRS; Posner et al., 2011) serves as the outcome measure, which assesses the constructs of suicidal behavior (i.e., actual, aborted, or interrupted attempts), severity, and lethality. Although suicidal behavior is the primary outcome of interest, suicidal ideation (passive, active, intensity) will also be assessed by the C-SSRS. The C-SSRS has four constructs relevant to recent suicidal ideation (SI): 1) severity (1=wish to be dead, 2=nonspecific active suicidal thoughts, 3=suicidal thoughts with methods, 4=suicidal intent, and 5=suicidal intent with plan); 2) intensity (sum across six items each rated 0 to 5: most severe ideation, frequency, duration, controllability, deterrents, and reason); 3) behavior; and 4) lethality.

OTHER OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item measure designed to identify individuals whose alcohol use places them at risk for alcohol-related problems, or who are actually experiencing such problems. The AUDIT assesses frequency of drinking, dependence symptoms, and signs of harmful consumption, each on a four point scale, providing a total score between 0 and 40. A score of 0 indicates that the respondent has never had problems from alcohol, sores of 1 to 7 indicate low-risk consumption of alcohol, scores of 8 to 14 suggest harmful consumption of alcohol, and scores of 15 or more indicate moderate-severe alcohol use disorder.
Beck Scale for Suicide Ideation (BSS) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The BSS is a 21-item self-report instrument assessing individual's thoughts, attitudes and intentions regarding suicide over the past week, including attitudes toward living and dying, expected reactions to these thoughts, and frequency of past suicidal behavior.The items provide participants with three response options (e.g., "I have no wish to die", "I have a weak wish to die", or "I have a moderate to strong wish to die") and are rated on a scale from 0 to 2, based on intensity. Scores are summed to provide a total score indicative of suicide risk. A higher score indicates a higher risk.
The Beck Depression Inventory-II (BDI-II) | Pre-intervention, Post-intervention (Up to six weeks)
  The BDI-II is a 21-item self-report measure of the severity of depressive symptoms. The items are scored from 0 to 3 to assess the level of symptom severity. Responses on the items are summed to derive a total scale score, with higher scores suggestive of higher depressive symptom severity.
Altman Self-Rating Mania Scale (ASRM) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The ASRM is a self-administered five-item questionnaire regarding mania/hypomania. Each item is rated on a five-point anchored Likert scale, generating total scale scores ranging from 0 to 20. A total score of greater than or equal to 6 indicates symptoms of mania/hypomania.
World Health Organization Quality of Life-Brief (WHOQOL-BREF) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The WHOQOL-BREF is an abbreviated 26-item quality of life assessment. It produces scores for four domains of quality of life, namely, physical health, psychological health, social relationships and environment. Higher scores indicate greater satisfaction with life or health and higher quality of life.
Impulsive/Premeditated Aggression Scale (IPAS) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The IPAS is a fifteen item questionnaire that assesses impulsive aggression and premeditated aggression. Participants are asked to indicate how much each item characterized a past incident of aggression during the last 6 months and complete the IPAS in relation to those acts on a 5-point Likert scale from strongly agree to strongly disagree. High scores are indicative of greater aggression.
Interpersonal Needs Questionnaire-15 (INQ-15) Score | Pre-intervention, Post-intervention (Up to six weeks)
  The INQ- 15 is a measure of perceived burdensomeness and belongingness. All statements are rated on a 7-point scale from 1 (not at all true for me) to 7 (very true for me), with higher summed scores corresponding to higher levels of perceived burdensomeness and belongingness.
Acquired Capability for Suicide Scale (ACSS) Score | Post-intervention (Up to six weeks)
  The ACSS is a 7-item self-report instrument designed to assess levels of acquired capability. On each item, participants are asked to report how much they identify with the item, using a 5-point Likert-scale ranging from 0 "Not at All Like Me" to 4 "Very Much Like Me." Total scores may range from 0 to 28, with higher scores indicating greater levels of acquired capability.
Psychache Scale Score | Post-intervention (Up to six weeks)
  The Psychache Scale is a 13- item self-report scale of psychological pain using a 5-point Likert scale. A higher score is predictive of suicidal ideation beyond the influence of depression and hopelessness.

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Lamis, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Au JS, Martinez de Andino A, Mekawi Y, Silverstein MW, Lamis DA. Latent class analysis of bipolar disorder symptoms and suicidal ideation and behaviors. Bipolar Disord. 2021 Mar;23(2):186-195. doi: 10.1111/bdi.12967. Epub 2020 Jul 8. PMID 32579284